CLINICAL TRIAL: NCT03378544
Title: Engaging Traditional Birth Attendants to Reduce Maternal Depression in Rural Kenya
Acronym: ENGAGE-TBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Africa Institute of Mental and Brain Health (AFRIMEB) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AfricaMHF
Record Dates: First submitted 2017-12-05; First posted 2017-12-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Patients with suicidal ideation and depression will receive psychosocial interventions adapted from the WHO mental health Global Action Programme Intervention Guide (mhGAP-IG). The intervention will involve psycho-education to patients on the importance of maintaining interest in activities that they used to do, regular sleep cycles, physical activity and social activity.
  Interventions: Behavioral: mhGAP
- Control group (No Intervention): Patients with suicidal ideation and depression will be trained on how to refer patients suffering from depression, using a referral note to the nearest health centre for further treatment

INTERVENTIONS:
Behavioral: mhGAP — The intervention will involve psycho-education to patients on the importance of maintaining interest in activities that they used to do, regular sleep cycles, physical activity and social activity
  Arms: Experimental arm

SUMMARY:
Evidence from Low and Middle Income Countries has demonstrated the effectiveness of various psychosocial approaches for depression. However, there are no mental health specialists to deliver these interventions especially in rural African settings. This study aims at testing the effectiveness of mental health Global Action Programme (mhGAP-IG) psychosocial interventions among Traditional Birth Attendants (TBAs) for pregnant mothers. The outcomes of this intervention will result into depression reduction in the mothers that will lead to better care during pregnancy and for their infants, allowing for long-term impact on their physical and the psychological wellbeing and that of their children.

DETAILED DESCRIPTION:
Evidence from Low and Middle Income Countries has demonstrated the effectiveness of various psychosocial approaches for depression. However, there are no mental health specialists to deliver these interventions especially in rural African settings. This study aims at testing the effectiveness of mental health Global Action Programme (mhGAP-IG) psychosocial interventions among Traditional Birth Attendants (TBAs) for pregnant mothers seeking the services of TBAs and suffering from maternal depression.

A cluster randomized controlled trial with two sub-counties in Makueni County (rural Kenya) as the clusters, randomized into either intervention or control arms will be used. TBAs in the intervention arm will receive training on mhGAP-IG while those in the control arm will only be requested to refer patients to nearest clinics and continue with their routine care, except in circumstances of pregnancy-related complications or severe medical conditions. All pregnant mothers will be eligible for inclusion.

Qualitative measures will be used to explore community and other stakeholder views regarding the integration of TBAs into mental health care and promoting dialogue with the formal health sector. Various questionnaires will be administered at 0, 3, 6 and 9 months in order to test the effectiveness of the intervention at various intervals. Interviews will be conducted at 9 months for randomly selected mothers receiving the intervention and those in the control arm, for purposes of describing and evaluating their experiences regarding use of TBA and health care workers' services. The survival and physical wellbeing of the baby will also be measured using the labour process, birth and subsequent weight of the baby, completed schedules of immunization and developmental milestones until 6 months.

The outcomes of this intervention will result into depression reduction in the mothers that will lead to better care during pregnancy and for their infants, allowing for long-term impact on their physical and the psychological wellbeing and that of their children.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of between 16 and 26 weeks
* A positive score on EPDS
* Confirmed diagnosis of depression using the Mini International Psychiatric Interview
* Provision of an informed consent

Exclusion Criteria:

* Actively suicidal
* Severe mental disorders and/or medical conditions requiring immediate medical attention
* A negative score on EPDS
* Pregnancy-related complications
* Decline to provide informed consent

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant mothers seeking the services of traditional birth attendants
Enrollment: 220 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | 0, 3, 6, and 9 months
  The proportion of patients (mothers with maternal depression) with reduction of depressive symptoms at 3, 6, and 9 months from baseline, using the Edinburgh Postnatal Depression Scale. This tool has adequate sensitivity and specificity to identify depressive symptoms in the antenatal and postnatal periods. A score is calculated by adding the individual items for each question. A total score of 11 or more in the Kenyan context is considered a flag for the need for follow up of possible depressive symptoms.

SECONDARY OUTCOMES:
Intimate Partner violence | Baseline
  The proportion of depressed patients at the TBA clinics experiencing intimate partner violence using the World Health Organization instrument to measure partner violence. This questionnaire measures violence from various aspects such as (i) physical, sexual, emotional, controlling behaviours and physical violence in pregnancy; (ii) physical and forms of violence by non-partners since age 15 years and (iii) Childhood sexual abuse before age 15 years. A "yes" in any of the items in the specific forms of violence indicates a positive score for that type of violence.
Quality of life of mothers with depression | 0, 3, 6, and 9 months
  Change from baseline to 3, 6, and 9 months in quality of life domains using the World Health Organization Quality of Life questionnaire. The minimum and maximum scores for physical, psychological, social and environmental domains are (7-35), (6-30), (3-15) and (8-40) respectively. The domains are scored through a simple algebraic summation of each item in that scale and the raw scores transformed into a 0-100 scale by subtracting lowest possible raw score from actual raw score and dividing the total by the possible raw score range, then the total is multiplied by 100. Higher scores on each of the domains indicate higher quality of life.
Satisfaction levels | 0, 3, 6, and 9 months
  Change in satisfaction levels among patients seeking TBA services
Suicidality | 0, 3, 6, and 9 months
  The proportion of patients with reduced suicidal behaviors such as ideations or attempts as measured using the Beck's Suicidality Scale at 3, 6, and 9 months. This scale assesses a patient's thoughts, plans and intent to commit suicide. There are no specific cut-off scores for severity classification. Therefore, the total scores calculated through summation of the items range from 0 to 42. Increasing scores reflect greater suicide risk.
Disability | 0, 6, and 9 months
  Change from baseline to 6, and 9 months in disability scores using the World Health Organization Disability Assessment Schedule. This scale asks difficulties related to health/mental conditions. The "item-response-theory" (IRT)-based scoring which takes into account multiple levels of difficulty for each item is used. After summing the scores for all six different functioning domains: cognition, mobility, self-care, getting along, life activities (household and work/school) and participation, the summary scores are converted into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability). High scores on a particular domain indicate significant and problematic areas for the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Christine W Musyimi, Principal Investigator — Africa Institute of Mental and Brain Health (AFRIMEB)
Locations (1):
- Tawa and Kanzokea, Makueni Boma, Makueni County, Kenya

IPD SHARING:
Plan to Share IPD: No